CLINICAL TRIAL: NCT05553912
Title: QBSafe: a Randomized Trial of a Novel Intervention to Improve Care for People Living With Type 2 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000032654; 1R01DK129616-01A1 (NIH)
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Type2Diabetes; Diabetes
Keywords: A1c; HbA1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized clinical trial of usual care with a behavioral intervention (use of conversation cards during routine clinical encounters) compared with usual care alone. The study will randomize 10-15 clinicians and 72 of their patients with type 2 diabetes to each arm. Data collected includes medical record data, patient and clinician surveys, and audio-visual recordings of clinical encounters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QBSafe intervention (Experimental)
  Interventions: Behavioral: QBSafe
- usual care (No Intervention)

INTERVENTIONS:
Behavioral: QBSafe — an intervention comprised of (a) a set of conversation cards (QBSafe ASK) designed to enable patients to identify aspects of life with diabetes important to them and to share them with their clinician to obtain their input; and (b) materials that help clinicians respond to patient concerns.
  Arms: QBSafe intervention

SUMMARY:
Glycemic control is often the main indicator of successful diabetes care, but a singular focus on glycemic control may lead to patients' overall health and wellbeing being overlooked or undervalued. The investigators have previously developed an intervention comprised of (a) a set of conversation cards designed to enable patients to identify aspects of life with diabetes important to them and to share them with their clinician to obtain their input; and (b) materials that help clinicians respond to patient concerns. The investigators will now conduct a randomized clinical trial to test the feasibility of the research procedures and efficacy of the intervention with respect to patient reported outcome measures.

DETAILED DESCRIPTION:
The goal of this study is to assess the feasibility and efficacy of usual care with the QBSafe intervention compared to usual care alone within a cluster randomized clinical trial among patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Clinicians

* any physicians, residents, nurse practitioners, and physician assistants who participate in the care of patients with type 2 diabetes (DM2) management (DM2) and prescribe medications for them

Participants

* diagnosed with DM2
* able to sign informed consent
* fluent in either English or Spanish
* HbA1c >8%

Exclusion Criteria:

* Participants for whom an HbA1c target >8% is clinically reasonable (e.g., those with limited life expectancy) and/or aligned with goals/preferences

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Illness intrusiveness measured by the Illness Intrusiveness Ratings Scale (IIRS) at Month 6 | Month 6
  The change in illness intrusiveness measured by the validated Illness Intrusiveness Ratings Scale (IIRS). IIRS is comprised of 13 items that ask participants to rate the degree to which their "illness and/or its treatment" interfere with life domains central to quality of life. the score is calculated by summing the 13 items creating a value between 13 to 91, where higher scores indicate increased illness intrusiveness. Analysis will assess the 6 months response as the outcome adjusting for arm and the initial score
HbA1c at Month 6 | Month 6
  HbA1c value at month 6. Analysis will model the 6 month HbA1c assessment adjusting for arm and the initial score.

SECONDARY OUTCOMES:
Diabetes distress will be measured using the Diabetes Distress Scale (DDS-17) at Month 6 | Month 6
  The DDS is a validated 17-item self-report instrument where each item is rated on a 6-point Likert scale from (0) "not a problem" to (6) "a serious problem." The scale yields a total DDS score, plus scores for 4 subscales: emotional burden, regimen distress, physician distress, and interpersonal distress. Total and subscale scores are calculated using mean item scores, which are then categorized as little or no distress (< 2.0), moderate distress (greater than or equal to 2.0 and less than or equal to 2.9) and high distress (greater than equal to 3.0). Moderate and high distress are considered 'clinically significant.'
Treatment burden will be assessed using the Treatment Burden Questionnaire (TBQ) at Month 6 | Month 6
  The TBQ is a self-reported questionnaire assessing the burden of treatment without restricting its scope to a single condition or treatment context. It is composed of 15 items rated on a Likert scale ranging from 0 (no impact) to 10 (considerable impact) related to the burden associated with taking medicine, self-monitoring, laboratory tests, physician visits, need for organization, administrative tasks, following advice on diet and physical activity, and social impact of the treatment. Item scores can be summed into a global score, ranging from 0 to 150. Higher scores reflect higher treatment burden.
Quality of life was assessed using the Visual Analogue Scale (VAS) at Month 6. | Month 6
  To assess global quality of life, a single-item VAS survey will be used with scale ranging from 0 (worst possible)-to-100 (best possible).
Hypoglycemia measured at month 6 | Month 6
  Hypoglycemia will be measured by asking participants about the frequency of any hypoglycemia (defined by a glucose level below 70 mg/dl [Level 1 hypoglycemia] or symptoms consistent with hypoglycemia), any blood glucose level below 54 mg/dl (Level 2 severe hypoglycemia), or any hypoglycemia requiring assistance from another person to treat.
Quality of communication assessed using 3 questions from the CAHPS Clinician and Group survey | up to 6 months
  The quality of communication will be assessed with a modified version of 3 questions from the CAHPS Clinician and Group survey. These questions indicate the extent to which the communication is patient-centered, covering technical (explain things in a way you could understand) and affective (show respect for what you have to say) communication.

OTHER OUTCOMES:
Patient satisfaction survey | up to 6 months
  Patients will rate their satisfaction with the approach used during the encounter on a 5-point Likert scale, which could have been usual care alone or usual care with the QBSafe ASK.
Clinician satisfaction survey | up to 6 months
  Clinicians will rate their satisfaction with the approach used during the encounter on a 5-point Likert scale, which could have been usual care alone or usual care with the QBSafe ASK.

CONTACTS AND LOCATIONS:
Overall Officials: Kasia Lipska, MD MHS, Principal Investigator — Yale University
Locations (1):
- Fair Haven Community Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes